CLINICAL TRIAL: NCT02345837
Title: Effect of Local Endometrial Injury on Pregnancy Outcomes During Ovulation Induction Cycles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al Hayat National Hospital (Other)
Collaborators: Menoufia University (Other)
Responsible Party: Principal Investigator, mohamed maher, assisstant professor, Al Hayat National Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: menoufia ob/gyn
Record Dates: First submitted 2015-01-20; First posted 2015-01-26 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Asymptomatic Diseases
MeSH Terms: conditions — Asymptomatic Diseases | interventions — Clomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clomiphene and endometrial sampling (Active Comparator): Couples who will undergo endometrial sampling in the luteal phase of the cycle preceding ovulation induction by clomiphene citrate.
  Interventions: Device: endometrial sampling; Drug: clomiphene citrate
- clomiphene citrate (Active Comparator): Couples who will undergo ovulation induction with clomiphene citrate.
  Interventions: Drug: clomiphene citrate

INTERVENTIONS:
Device: endometrial sampling — injury to the endometrium
  Arms: clomiphene and endometrial sampling
Drug: clomiphene citrate — ovulation induction by 100mg clomiphene citrate
  Other Names: clomid

SUMMARY:
The aim of this study is to detect whether or not performing an endometrial sampling in the cycle preceding ovulation induction with clomiphene citrate can improve pregnancy outcomes in the next cycle.

DETAILED DESCRIPTION:
Patients will be randomized using a list of computer generated random sample into two groups:

Group 1: Couples who will undergo endometrial sampling in the luteal phase of the cycle preceding ovulation induction by clomiphene citrate.

Group 2: Couples who will undergo ovulation induction with clomiphene citrate. The drug chosen for ovulation induction in both groups will be clomephine citrate.

Timing and technique of endometrial sampling:

Timing: from day 15 to day 24 of the cycle preceding ovulation induction cycle. Technique: this will be done using the pipelle method (Williams et al., 2008).

The procedure is as follows:

1. Vaginal speculum to expose the uterine cervix then sterilization by saline.
2. The piston positioned at the extreme distal end of the sheath then the Pipelle is inserted gently through the cervical canal into the cavity of the uterus.
3. While holding the sheath in position with one hand, the other hand rapidly pulls the piston firmly and without interruption.
4. A negative pressure within the sheath will draw the tissue into the curette opening at the distal end of the sheath and captures the separated tissue within its lumen.

ELIGIBILITY:
Inclusion Criteria:

1. Male partner should have a normal semen count and motility according to world health organization criteria (Murray et al., 2012).
2. Primary, secondary or unexplained infertility for at least one year.
3. Failure to conceive with clomiphene citrate in spite of good follicular response for at least 3 cycles.
4. Age varies from 20-35 years with at least one year of infertility.
5. Body mass index between 19-30 kg/m2.
6. Day 2 serum FSH< 12 IU/ml.
7. Normal uterine cavity on hystrosalpingography.
8. At least one patent tube of normal appearance on HSG.
9. No previous attempts of intrauterine insemination (IUI) or in vitro fertilization (IVF).

Exclusion Criteria:

1. Infertility due to tubal factor or male factor.
2. Intrauterine organic pathology (myoma, polyp, adhesions) by hystrosalpingogram or diagnostic hysteroscope.
3. Hypogonadotrophic hypogonadism.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate. | one year
Miscarriage rate. | one year
Multiple pregnancy rates | one year

CONTACTS AND LOCATIONS:
Overall Officials: menoufia university, Study Chair — menoufia fuculty of medicine
Locations (1):
- Menoufia University, Shebin Elkom, Egypt

REFERENCES:
- [Derived] Helmy MEE, Maher MA, Elkhouly NI, Ramzy M. A randomized trial of local endometrial injury during ovulation induction cycles. Int J Gynaecol Obstet. 2017 Jul;138(1):47-52. doi: 10.1002/ijgo.12178. Epub 2017 May 4. PMID 28397981